CLINICAL TRIAL: NCT03944447
Title: Outcomes Mandate National Integration With Cannabis as Medicine
Acronym: OMNI-Can
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: OMNI Medical Services, LLC (Network)
Collaborators: OMNI Medical Services Inc (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00033337
Record Dates: First submitted 2019-05-03; First posted 2019-05-09 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-02

CONDITIONS: Chronic Pain; Chronic Pain Syndrome; Chronic Pain Due to Injury; Chronic Pain Due to Trauma; Fibromyalgia; Seizures; Hepatitis C; Cancer; Crohn Disease; HIV/AIDS; Multiple Sclerosis; Traumatic Brain Injury; Sickle Cell Disease; Post Traumatic Stress Disorder; Tourette Syndrome; Ulcerative Colitis; Glaucoma; Epilepsy; Inflammatory Bowel Diseases; Parkinson Disease; Amyotrophic Lateral Sclerosis; Chronic Traumatic Encephalopathy; Anxiety; Depression; Insomnia; Autism; Opioid-use Disorder; Bipolar Disorder; Covid19; SARS-CoV Infection; COVID-19; Corona Virus Infection; Coronavirus
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Seizures; Hepatitis C; Neoplasms; Crohn Disease; Acquired Immunodeficiency Syndrome; Multiple Sclerosis; Brain Injuries, Traumatic; Anemia, Sickle Cell; Stress Disorders, Post-Traumatic; Tourette Syndrome; Colitis, Ulcerative; Glaucoma; Epilepsy; Inflammatory Bowel Diseases; Parkinson Disease; Amyotrophic Lateral Sclerosis; Chronic Traumatic Encephalopathy; Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders; Autistic Disorder; Opioid-Related Disorders; Bipolar Disorder; COVID-19; Severe Acute Respiratory Syndrome; Coronavirus Infections | interventions — Medical Marijuana

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cannabis users (Experimental): Most patients will have used cannabis before their initial physician visit, and many current patients will be returning for an in-person follow-up. Patients will be given the survey shortly after the physician encounter to assess baseline parameters with current cannabis use. Any patient who is "cannabis-naïve", defined as no use within the past year or longer, will be placed into a separate data analysis arm. The investigators will follow up with patients again at 3, 6, 9, and 12 months with the online survey. Patients returning for their annual physician encounter will continue on the 3-month survey schedule until the end of the study, or if lost to follow-up. There may be slight variations in the interval based on state law, for example in Florida the in-person follow-up with the physician is required every 210 days, and some states allow for 2 year in-person visits. Every attempt will be made to adhere to a 3-month interval survey distribution.
  Interventions: Drug: Cannabis, Medical; Device: RYAH-Medtech Inhaler
- Cancer prevention (Experimental): Non-cancer patient medical cannabis users with extensive or life-long cannabis use will be compared to the general population for incidence and prevalence of development of cancer. The hypothesis is that cannabis use acts as a cancer preventive substance.
  Interventions: Drug: Cannabis, Medical; Device: RYAH-Medtech Inhaler
- Life-Threatening Conditions (Experimental): Opioids are a class of drugs naturally found in the opium poppy plant. Opioids are often used as medicines because they contain chemicals that relax the body and can relieve pain. Prescription opioids are used mostly to treat moderate to severe pain. Opioids can also make people feel very relaxed and "high" - which is why they are sometimes used for non-medical reasons. This can be dangerous because opioids can be highly addictive, and overdoses and death are common.
  From 1999 to 2017, more than 700,000 people have died from a drug overdose. Around 68% of the more than 70,200 drug overdose deaths in 2017 involved an opioid.
  In 2017, the number of overdose deaths involving opioids was 6 times higher than in 1999.
  On average, 130 Americans die every day from an opioid overdose.
  This study will focus on examining outcomes of patients that have been treated with cannabis as a replacement or alternative to life-threatening opioids or other prescription drugs.
  Interventions: Drug: Cannabis, Medical; Device: RYAH-Medtech Inhaler
- COVID-19 / SARS-CoV-2 (Experimental): Inhibition of viral entry and thereby spread constitute plausible therapeutic avenues. Similar to other respiratory pathogens, SARS-CoV2 is transmitted through respiratory droplets, with potential for aerosol and contact spread. It uses receptor-mediated entry into the human host via angiotensin-converting enzyme II (ACE2) that is expressed in lung tissue, as well as oral and nasal mucosa. Modulation of ACE2 levels in these gateway tissues may prove a plausible strategy for decreasing disease susceptibility. Cannabis sativa, especially one high in the anti-inflammatory cannabinoid cannabidiol (CBD), has been proposed to modulate gene expression and inflammation and possess anti-cancer and anti-inflammatory properties. Covid-19 infection rates in cannabis users will be compared to rates in the general population. Severity of persistent symptoms in cannabis users testing positive for active infection and/or antibodies will also be compared to the general population.
  Interventions: Drug: Cannabis, Medical; Device: RYAH-Medtech Inhaler

INTERVENTIONS:
Drug: Cannabis, Medical — Patients will be given medical cannabis recommendations and certifications commensurate with the state law in which the encounter occurs. The variations in mechanisms between the states for recommending, registering, certifying, and developing mandated treatment plans or doses will be adhered to; however, variations in state law and cannabis programs should not cause variation in the study design because the end-result is still the same with patients being treated with medical cannabis.
  Other Names: Marijuana Medical; Marijuana Treatment
Device: RYAH-Medtech Inhaler — Our research study will involve incorporation of RYAH-Medtech company's devices into our protocols. They have an inhaler and a transdermal patch for both hemp-derived CBD and cannabis. RYAH has developed an integrated phone app for tracking product use and patient response. They are currently involved in clinical trials in Europe. OMNI Medical will integrate the partner with RYAH device for several reasons. Primary goals will involve using their integrated smart phone app to collect and secure large quantities of data. Secondary goals will include FDA approval as a medical device. The specific cannabis strain will be tracked using scannable QR codes programed into the smart phone app. This will allow us to track patient feedback and capture data on usage. OMNI Medical will have patients use RYAH's products as part of and FDA Investigational Device Exemption, which requires an IRB. Use of the devices would be completely voluntary by study participants.

SUMMARY:
This will be a multistate, multicenter clinical study to determine the efficacy and safety of medical cannabis for a wide variety of chronic medical conditions.

DETAILED DESCRIPTION:
Medical cannabis has been legal in parts of the USA since 1996, with the stated intention of reducing pain (both acute and chronic) as well as for treatment of multiple other conditions. The original implementation of medical cannabis in the USA was implemented in California as a compassionate measure to treat the HIV/AIDS epidemic. Additional studies have shown promising outcome for patients with multiple sclerosis, seizures, cancer, and other chronic conditions. However, there have been few comprehensive studies that have actually measured whether cannabis is an effective treatment for pain reduction. There is an absence of multistate, multicenter clinical studies with cannabis as medicine, not only in the USA but globally. With the expansion of medical cannabis into more than 38 states in the US, this type of clinical study is now feasible.

On March 11, 2020, the World Health Organization formally characterized coronavirus, COVID-19, as a global pandemic and health systems globally are continuing their efforts to manage the outbreak. Coronavirus disease COVID-19 is an infectious disease caused by a newly discovered coronavirus. With the rapidly growing pandemic of COVID-19 caused by the new and challenging to treat zoonotic SARS-CoV2 coronavirus, there is an urgent need for new therapies and prevention strategies that can help curtail disease spread and reduce mortality. Inhibition of viral entry and thereby spread constitute plausible therapeutic avenues.

This study will utilize an anonymous novel online questionnaire to determine study participants' qualifying condition(s) for medical cannabis use, cannabis ingestion method, frequency of use, prescription drug use, and demographic information. Secondary factors will include evaluation of pain control, quality of life metrics, any adverse side effects from cannabis use, as well as changes in adjunctive treatments. Patients will be given medical cannabis recommendations and certifications commensurate with the state law in which the encounter occurs. The variations in mechanisms between the states for recommending, registering, certifying, and developing mandated treatment plans or doses will be adhered to; however, variations in state law and cannabis programs should not cause variation in the study design because the end-result is still the same with patients being treated with medical cannabis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a Qualifying Condition for Medical Marijuana
* Must be 18 years or older unless they have consent from their parent or legal guardian as defined under state law parameters
* Must be willing to complete online surveys at baseline and the follow up points in this study

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Inability to provide informed consent
* Inability to complete study visits or questionnaires
* Active suicidality or psychosis, that could be exacerbated by the administration of cannabis

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevention of COVID-19 | Five years
  Covid-19 infection rates in cannabis users will be compared to rates in the general population. Our online questionnaire responses will compare infection rates of cannabis users in this study against the Johns Hopkins University Coronavirus Research Center data (https://coronavirus.jhu.edu).
Treatment of COVID-19 | Five years
  Severity of persistent symptoms in cannabis users testing positive for active infection and/or antibodies will also be compared to the general population. Patients will answer the widely used FLU-PRO questionnaire, which asks about flu symptoms and severity, to capture diagnoses, symptoms, and medical interventions related to COVID-19. The data from cannabis user patients will be compared with national and international data surveys, such as the Covid Symptom Study (https://covid.joinzoe.com/us-2).
Treatment of Symptoms | Five years
  The primary objective is to assess the efficacy and safety of medical cannabis as medicine for treatment of chronic pain and other chronic debilitating diseases. Pain will be measured by Brief Pain Inventory (BPI) numeric scale. Change from baseline in BPI will be assessed at 3-month intervals. For prospective associations between cannabis use and outcomes, use of a lagged mixed-effects models will examine temporal associations between cannabis use and pain severity, opioid sparing, and patient satisfaction. Data will be analyzed from baseline and the annual follow-up waves.

SECONDARY OUTCOMES:
Cannabis Impact on Quality of Life | Five years
  Secondary objectives include evaluating increases or decreases in quality of life, and increases or decreases in concomitant opioid use. Satisfaction with treatment will be measured by a Visual Analog Score (VAS). Change From baseline in Satisfaction with treatment measured by (VAS) be assessed at 3-month intervals.
Cannabis Route and Dosing | Five years
  Tertiary objectives will examine preferences for routes of administration, and preferences for THC / CBD ratios. Categorical factors will be summarized using frequencies and percentages, while continuous measure distributions will be described using means, standard deviations, and quartiles of interest.
Monitoring Adverse Events | Five years
  Incidence of Treatment-Related Adverse Events will be measured by Physician Global Assessment (PGA) numeric scale. Number of participants with Treatment-Related Adverse Events will be assessed by CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ryan O Lakin, MD JD, Principal Investigator — OMNI Medical Services Inc
Locations (16):
- United States (16):
  - OMNI Medical Services, Boca Raton, Florida
  - OMNI Medical Services, Bradenton, Florida
  - OMNI Medical Services, Fort Lauderdale, Florida
  - OMNI Medical Services, Fort Myers, Florida
  - OMNI Medical Services, Gainesville, Florida
  - OMNI Medical Services, Merritt Island, Florida
  - OMNI Medical Services, Miami, Florida
  - OMNI Medical Services, Ocoee, Florida
  - OMNI Medical Services, Pensacola, Florida
  - OMNI Medical Services, Pompano Beach, Florida
  - OMNI Medical Services, Tampa, Florida
  - OMNI Medical Services, Wesley Chapel, Florida
  - OMNI Medical Services, Beechwood, Ohio
  - OMNI Medical Services, Bowling Green, Ohio
  - OMNI Medical Services, Sandusky, Ohio
  - OMNI Medical Services, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: OMNI Medical Services Website — http://omnidoctors.com/